CLINICAL TRIAL: NCT00302653
Title: Program of Rasburicase in the Treatment of Hyperuricemia in Children and Adolescent Patients With or at Risk of Tumor Lysis Syndrome.
Brief Title: Rasburicase in Tumor Lysis Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: L_9436
Record Dates: First submitted 2006-03-10; First posted 2006-03-14 (Estimated); Last update posted 2009-09-25 (Estimated); Status verified 2009-09

CONDITIONS: Hyperuricemia
MeSH Terms: conditions — Hyperuricemia | interventions — rasburicase

ARMS (1):
- 1 (Experimental): Rasburicase 0,20mg/Kg/Day once a day 3-7 days
  Interventions: Drug: Rasburicase

INTERVENTIONS:
Drug: Rasburicase — Rasburicase 0,20mg/Kg/Day once a day 3-7 days

SUMMARY:
The purpose of this study is to determine whether rasburicase is effective and safety in correcting hyperuricemia.

ELIGIBILITY:
List of inclusion Criteria:

* Acute hyperuricemia patients(uric acid>8.0 mg/dl) before/during chemotherapy for hematologic malignancies.

List of exclusion Criteria:

* Hypersensitivity to uricases or any of the excipients.
* Known history of hemolytic anemia (G6PD deficiency).

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 33 (Actual)
Dates: Start 2006-02; Primary Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with uric acid greater-than-normal laboratory levels (hyperuricemia) | 24-48 hours after last dose of rasburicase
Percentage of patients with uric acid greater-than-normal laboratory levels (hyperuricemia) | 28 (+- 3) days after the last dose of rasburicase
Adverse events occurrence | During the study

CONTACTS AND LOCATIONS:
Overall Officials: Jaderson Lima, Study Director — Sanofi-aventis administrative office Brazil
Locations (1):
- Sanofi-aventis administrative office, São Paulo, Brazil